CLINICAL TRIAL: NCT05853926
Title: Spinal Manipulation With Laser Therapy Versus Dry Needling in Chronic Lower Backache: Randomized Controlled Trial
Brief Title: Spinal Manipulation With Laser Therapy Versus Dry Needling in Chronic Lower Backache
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPT/Batch-Fall18/530
Record Dates: First submitted 2023-03-18; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spinal Manipulation With Laser Therapy (Experimental)
  Interventions: Diagnostic Test: Spinal Manipulation With Laser Therapy
- Dry Needling (Other)
  Interventions: Diagnostic Test: Dry Needling

INTERVENTIONS:
Diagnostic Test: Spinal Manipulation With Laser Therapy — Spinal Manipulation With Laser Therapy in Chronic Lower Backache
  Arms: Spinal Manipulation With Laser Therapy
Diagnostic Test: Dry Needling — Dry Needling in Chronic Lower Backache
  Arms: Dry Needling

SUMMARY:
To determine the effectiveness of spinal manipulation with laser therapy versus dry needling for pain, disability and fear of movement in chronic low backache

ELIGIBILITY:
Inclusion Criteria:

* Those patients will be included in the study who have chronic low back pain (12 week duration).

both genders aged 18-60 years low back pain

Exclusion Criteria:

* Those patients will be excluded in the study who have needle phobia, any infection, cancer, dermal changings, heart transplant, pregnancy, rheumatic fever(25)fracture, cauda equina syndrome, arrhythmia, sensory deficiency, mental illness, surgery, osteoporosis, low term use of steroid

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index scale | 6 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Chaudary Muhammad Akram Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No